CLINICAL TRIAL: NCT02122601
Title: An Open-label, Single Arm, Multi-center, Phase 3 Study to Evaluate the Safety and Efficacy of Retreatment With Intra-articular LBSA0103 Injections in the Patients With Osteoarthritis of the Knee
Brief Title: A Clinical Trial to Evaluate the Safety and Efficacy of Retreatment With Intra-articular LBSA0103 Injections in the Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LG-HACL013
Record Dates: First submitted 2014-04-16; First posted 2014-04-24 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee

ARMS (1):
- LBSA0103 (Other): single arm , LBSA0103 only
  Interventions: Drug: LBSA0103 (BDDE cross-linked sodium hyaluronate gel)

INTERVENTIONS:
Drug: LBSA0103 (BDDE cross-linked sodium hyaluronate gel)

SUMMARY:
To assess the safety and efficacy of LBSA0103 (BDDE cross-linked sodium hyaluronate gel) when it is administered for the second time 26 weeks after its first administration in patients with osteoarthritis of the knee.

The Safety and efficacy of 26weeks after its first administration will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. A patient diagnosed with one or both knee osteoarthritis based on the clinical diagnosis criteria of the American College of Rheumatology (ACR) (there should be knee pain and in addition, at least three of the following six conditions have to be satisfied: 1. Over 50 years of age 2. Less than 30 minutes of morning stiffness 3. Crepitus on active motion 4 Bony tenderness 5. Bony enlargement 6. No palpable warmth of synovium)
2. Adult male and female patients of age 40 or above diagnosed with knee osteoarthritis with the Kellgren & Lawrence Grade of I - III by x-ray within 6 months before the screening visit (based on -2 weeks) or by x-ray at the screening visit
3. A patient who has at least one knee with a weight-bearing pain value of 40 mm or more when weight-bearing pain (100 mm-VAS) is measured
4. A patient taking aspirin at a low dose (300 mg or less per day) who is willing to take aspirin constantly at the same dose until the clinical study is completed and can refrain from taking aspirin within 24 hours before each visit.
5. A patient who can walk without depending on a walking aid such as walker, cane, etc. but if the patient has been using a walking aid on a daily basis from six months ago, the patient assessment can be conducted while including the walking aid and the walking aid must be used in the same way until the study is completed.
6. A patient who can understand the meanings of an efficacy measurement questionnaire well and complete it
7. A patient who heard an explanation about the purpose, method, effects, etc. of the clinical study and whose informed consent form has been signed by him/herself or subject's representative
8. A patient who falls under one of the following four cases

   * Patients who are surgically infertile
   * Post-menopausal women who are above 45 years of age and 2 years after the last menstruation
   * Fertile premenopausal female patients or male patients without having a surgical sterilization who have agreed to use at least two birth control methods (including one of barrier methods) for at least 13 weeks after the administration of the last investigational product to avoid pregnancy

     * Barrier methods: Condom, Diaphragm, Cervical cap(Pessary), Spermicide
     * Hormonal methods: Pills, Injection(Depot), Skin patch, Hormonal implant(Implanon), Vaginal ring
     * Intrauterine Devices(IUDs): Cooper IUD(Loop), Hormonal IUD(Mirena)
     * Natural methods: Basic body temperature, Ovulation period, Coitus interruptus, Abstinent
9. A patient who discontinued analgesics, NSAIDs, condroichin sulfate/glucosamine and physical therapy or oriental medical treatment (acupuncture, cubbing therapy, moxa treatment) within 2 weeks before the administration (washout period) and has a will to discontinue them from the screening visit of the study to the end (however, 300 mg less per day of aspirin and acetaminophen, a rescue therapy, can be taken)
10. A patient who didn't take any analgesic including aspirin and acetaminophen within 24 hours before the administration

Exclusion Criteria:

1. Body mass index > 32
2. A patient with rheumatoid arthritis, or other inflammatory or metabolic arthritis
3. A patient with infection or severe inflammation at the joint like septic arthritis
4. A patient with infection or skin disease at the site of administration
5. A patient with secondary knee osteoarthritis caused by ochronosis, hemochromatosis, systemic disease, etc.
6. A patient with a very painful musculoskeletal disease such as Sudek's atrophy, Paget's disease, or spinal disc herniation
7. A poly-artricular patient with a severe osteoarthritis symptom at other site (e.g., hip joint, etc.) which can have an effect on the assessment of the pain for knee joint
8. Patients diagnosed with knee osteoarthritis with the Kellgren & Lawrence Grade of IV in X-ray within 6 months before the screening visit (based on -2 weeks) or X-ray at the screening visit
9. A patient showing a clear loss in the joint space of patello-femoral joint (PFJ) in X-ray
10. A patient who took following drug before the administration of investigational product (baseline visit):

    * A patient who had HA at the target knee joint within the last 6 months
    * A patient who was given an intra-articular knee joint injection with steroidal agent within the last 3 months
    * A patient who used steroidal agent systemically by oral administration within the last 1 month (However, except for inhalant)
11. A patient with moderate to severe joint effusion which was found to be positive through patella tap test, etc.
12. A patient with alcoholism and alcoholic liver disease
13. A patient with a serious heart disease or hepatic and renal dysfunction or a patient who showed the following laboratory test value:

    * AST, ALT ≥ 3 times the upper limit of normal range
    * Serum creatinine > 2mg/dl
14. A patient who had a surgical procedure including arthroscopy on the target knee within the last 1 year (In case of a patient who had a history of joint surgery on other knee or hip joint, the patient shall be excluded if the assessment of the target knee is likely to be affected by that. )
15. A patient who has a history of knee replacement surgery on the target knee joint
16. A patient who does highly intensive aerobic exercise or heavy anaerobic exercise such as running or weight training which can have an effect on knee joint.
17. A patient who needs to use an anticoagulant agent concurrently (However, except for aspirin of 300 mg or less per day)
18. A patient who is mentally ill or can't understand the purpose and method of this clinical study
19. A patient who shows hypersensitivity reaction to the investigational product of this clinical study
20. A patient who is participating in other clinical study after having enrolled in this study, or participated in other clinical study within 1 month before the enrollment in this clinical study
21. A patient who is considered to have a difficulty undergoing the clinical study at the discretion of the Principal Investigator
22. A patient who was given one of the following drugs based on the day of administration:

    * A patient who was given anesthetic within the last 48 hours
    * A patient who took analgesics including acetaminophen and aspirin within the last 24 hour

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2014-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Adverse events for 13 weeks after the first and second administration | Week 13 from each baseline

SECONDARY OUTCOMES:
Local reactions at injection site after the first and second administration | Week 13 from each baseline
Adverse Events during total clinical study period | 0, 13, 26, 39 weeks
Vital signs | 0, 13, 26, 39 weeks
Laboratory exam | 0, 13, 26, 39 weeks
Change of Weight-bearing pain (100mm-VAS) from baseline | 0, 13, 26, 39 weeks
Change of WOMAC-likert assessment: Pain, Function, stiffness, Total score from baseline | 0, 13, 26, 39 weeks
Change of Patient Global Assessment (100mm-VAS) from baseline | 0, 13, 26, 39 weeks
Change of Investigator Global Assessment (100mm-VAS) from baseline | 0, 13, 26, 39 weeks
Change of rest pain(100mm-VAS) from baseline | 0, 13, 26, 39 weeks
Change of night pain(100mm-VAS) from baseline | 0, 13, 26, 39 weeks
Change of motion pain(100mm-VAS) from baseline | 0, 13, 26, 39 weeks
Physical assessment: swelling on knee joint, tenderness on pressure and the range of motion of knee joint | 0, 13, 26, 39 weeks
The Percentage of Subjects who took the Rescue Medicine (ACETAMINOPHEN REGIMEN) and Total Consumption | 0, 13, 26, 39 weeks
Responder Rate of subjects who showed a reduction by at least 20 mm or an improvement by at least 40% in the Weight-bearing pain (100 mmVAS) | 13, 26, 39 weeks
OMERACT-OARSI responder rate | 13, 26, 39 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea